CLINICAL TRIAL: NCT00009685
Title: Evaluation of an HIV-1 DNA Vaccine Encoding a Modified Gag-Pol Protein in Uninfected Adult Volunteers
Brief Title: HIV-1 Vaccine Test in Uninfected Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010079; 01-I-0079
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-03

CONDITIONS: Healthy; HIV Seronegativity
Keywords: Vaccine; HIV; Codon-Optimized; HIV Vaccine; Healthy Volunteer; HIV-1 DNA Vaccine; HIV Seronegativity; HIV Preventive Vaccine

INTERVENTIONS:
Drug: VRC4302

SUMMARY:
This study will test the safety of an experimental vaccine against HIV and will examine whether it causes an immune response to HIV virus proteins. A vaccine is given to try to create resistance or immunity to a disease or infection. The vaccine in this study is made from DNA (genetic material) of two HIV proteins called "gag" and "pol." Injected into a human, the viral DNA instructs the body to make small amounts of some HIV proteins. This study will see if the body then creates an immune response to these proteins. Study participants cannot catch HIV or AIDS from the DNA vaccine or proteins that may be made from it.

Healthy normal volunteers between 18 and 60 years of age may be eligible for this study. Candidates will provide a medical history, including information on sexual activity and drug use. They will have a physical examination, blood tests, urine test and chest X-ray. All candidates enrolled in the study must use a barrier method of contraception for sexual intercourse from the start of the study until 3 months after the last vaccination.

Participants will be assigned to one of two treatment groups: one will receive the experimental vaccine; the other will receive a control substance (inactive salt solution). The first five people assigned to the vaccine group will receive the lowest study dose of the vaccine. If this dose is safe, it will be increased three times for the next group of five and then eight times for the last group of five. Each group will have a total of seven people - five will receive the vaccine and two will get the salt solution.

Before the first injection, and possibly the second and third, a catheter (thin plastic tube) will be placed into a vein so that treatment can be given quickly if there is a reaction to the vaccine. Participants will receive three injections in an upper arm muscle-one injection a month for three months-with a needle-less device called a Biojector. For each injection, the volunteer will

* be observed for at least 1 hour after immunization
* record temperature and symptoms, including any effects at the injection site, for 2 days and report them to the clinic staff
* immediately report any side effects to a study physician or nurse.

Volunteers will have physical examinations and laboratory tests at certain times while they receive the vaccine and for a period afterwards. These procedures will require about 14 clinic visits of about 1 to 2 hours each, and up to 6 hours on vaccination days. Blood will be drawn at all visits. Some of the blood will be used for genetic tests, and some will be stored for future tests of the immune system and the body's response to the study vaccine. The study will last about 12 months from the date of the first injection. After it is completed, clinic staff may contact volunteers once or twice a year for at least 3 years to follow up.

DETAILED DESCRIPTION:
This is a Phase I randomized, controlled, double-blinded dose escalation study to examine toxicity, dose and immune response of an HIV plasmid DNA vaccine. The vector used in this study has been optimized for improved safety, expression and immunogenicity. We hypothesize that this vaccine will elicit immune responses to HIV. All work will be conducted at the National Institutes of Health.

Healthy, HIV-negative volunteers will be recruited and pre-screened to confirm that they meet all of the eligibility requirements for participation. Educational materials on DNA vaccines will be reviewed with and provided to participants before enrollment into the study. There will be 3 groups of 7 volunteers. Each group will receive a constant dose of the vaccine pGag(del fs)Pol delta PR delta RT delta IN/h (5 people) or a phosphate buffered saline (PBS) control (2 people) by intramuscular inoculation. Once safety has been established, successive groups will receive a higher dose. Study groups will receive three immunizations containing either 0.5 mg (Group 1), 1.5 mg (Group 2), or 4.0 mg (Group 3) of a DNA vaccine. Dose escalation will be initiated 5 weeks after the last volunteer in the previous dose group receives their first inoculation, providing there are no significant toxicities.

Vaccine-related adverse reactions will be evaluated at scheduled study visits and by study participant report. Immune response will be evaluated as described in Appendix II. Specimens to evaluate immunogenicity will be taken at baseline, and at the time points indicated in Appendix VIII. Unless contraindicated, subsequent inoculations using repeat plasmid vaccinations will be given 28 and 56 days after the first vaccinations. The estimated duration for each volunteer to complete immunizations and follow-up is 12 months.

ELIGIBILITY:
INCLUSION CRITERIA:

Participants must be between 18-60 years of age (no more than 10% of the volunteers to be over 50).

Male and female subjects are eligible. (For female participants: negative pregnancy test at the screening visit; for both male and female participants: agree to practice abstinence or use barrier contraception from the date of the first vaccination until 3 months after the final immunization.)

No significant findings on medical history, physical exam or screening lab studies as determined by clinic personnel

Willing to identify HIV infection risks and amenable to risk reduction counceling.

All subjects must understand the basis of transmission of HIV and agree to abstain from higher risk behavior for HIV infection.

Normal complete blood count and differential defined as:

Hematocrit greater than or equal to 34 percent for women and 38 percent for men; White blood cell count greater than or equal to 3,500/mm(3) and less than or equal to 10,000/mm(3) with no significant findings on differential; Total lymphocyte count greater than or equal to 800 cells/mm(3); Absolute CD4 count greater than or equal 400 cells/mm(3); Platelets 150,000-550,000 cells/cm(3).

Normal ALT and AST (less than or equal to 1.5 times institutional upper limit) and creatinine (less than or equal to 1.6 mg/dl).

Normal or low positive ANA titer (1 to 3 EU) if there is no clinical evidence of underlying disorders that are associated with a positive ANA, if no first degree relative has an autoimmune disease, and if anti-ENA antibodies are negative

Negative anti-dsDNA antibodies

Normal IgG levels

CPK less or equal to 2 times institutional upper limit

No significant findings on urinalysis

No significant findings on chest x-ray

Negative RPR (unless determined to be a false positive or a positive result is due to a prior-greater than 6 month-treated infection)

Negative for Hepatitis B surface antigen and anti-hepatitis C antibody

Negative for HIV by ELISA and DNA-PCR (below the limit of detection of the assay used) within 4 weeks of immunization (note that if a potential subject will not be allowed on study until further studies--potentially including repeat ELISAs, RT-PCR and DNA PCR--demonstrate that the subject is not infected with HIV)

Availability for follow-up for planned duration of the study (12 months)

Give informed consent by signing the Institutional Review Board (IRB) approved informed consent form(s)

Willingness to have samples stored and to have HLA testing

EXCLUSION CRITERIA:

History of immunodeficiency, chronic illness, malignancy, autoimmune disease, or use of immunosuppressive medications. Individuals with a history of cancer unless there has been surgical excision followed by a sufficient observation period to give a reasonable assurance of cure

Medical or psychiatric conditions which preclude subject compliance with the protocol.

Evidence of active drug or alcohol abuse

Tested positive to HIV at any time.

Live attenuated vaccines (including but not limited to measles, mumps, rubella and BCG) within 60 days of study (note: medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) are not exclusionary, but should be given at least 2 weeks away from HIV immunization)

Use of experimental agents within 30 days prior to study

Receipt of blood products or immunoglobulin in the past 6 months

Any history of anaphylaxis or history of other serious adverse reactions to vaccines

Prior receipt of HIV-1 vaccines

Pregnant or lactating women

Acute infectious illnesses within 1 month prior to initiation of immunization

History of splenectomy

Seizure disorder. A participant with a remote history (over 3 years) of seizure who have not received medications for 3 years or over are eligible if: 1. the seizures were febrile seizures under the age of 2; 2. secondary to alcohol withdrawal; or 3. it was a singular seizure.

Treatment with immunomodulators, except for NSAIDS, within 14 days prior to enrollment

Skin disease (e.g., eczema, psoriasis) affecting areas of immunization that precludes immunization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21
Dates: Start 2001-01; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Tighe H, Corr M, Roman M, Raz E. Gene vaccination: plasmid DNA is more than just a blueprint. Immunol Today. 1998 Feb;19(2):89-97. doi: 10.1016/s0167-5699(97)01201-2. No abstract available. PMID 9509764
- [Background] Fu TM, Ulmer JB, Caulfield MJ, Deck RR, Friedman A, Wang S, Liu X, Donnelly JJ, Liu MA. Priming of cytotoxic T lymphocytes by DNA vaccines: requirement for professional antigen presenting cells and evidence for antigen transfer from myocytes. Mol Med. 1997 Jun;3(6):362-71. PMID 9234241
- [Background] Ulmer JB, Deck RR, Dewitt CM, Donnhly JI, Liu MA. Generation of MHC class I-restricted cytotoxic T lymphocytes by expression of a viral protein in muscle cells: antigen presentation by non-muscle cells. Immunology. 1996 Sep;89(1):59-67. doi: 10.1046/j.1365-2567.1996.d01-718.x. PMID 8911141